CLINICAL TRIAL: NCT07086053
Title: Inter-rater And Intra-rater Reliability Of Biomechanical Skin Stiffness Characteristics Measurement Via MyotonPRO Device In Patients With Breast Cancer-Related Lymphedema (BCRL) And Their Relationship With Ultrasonographic Tissue Changes
Brief Title: Reliability of Myoton in Evaluating Skin Biomechanics in Breast Cancer-Related Lymphedema
Acronym: MYOLYMPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra Nur Turkmen, Lecturer / Specialist Physiotherapist, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FSM-MYOTON-2025-01
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer-Related Lymphedema
Keywords: Lymphedema; Breast Cancer; Myoton; Skin Stiffness; Ultrasound; Reliability
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group assignment. All participants will receive repeated MyotonPRO and ultrasound evaluations for skin biomechanical properties. No randomization or comparison between groups will be performed.
Masking Description: Although the study is single-arm, outcome assessments were performed by two blinded assessors to evaluate measurement reliability. No group assignment or treatment comparison is involved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphedema Assessment Group (Experimental): Patients with breast cancer-related lymphedema will undergo MyotonPRO and ultrasound measurements by two blinded raters to evaluate intra- and inter-rater reliability. No therapeutic intervention will be performed.
  Interventions: Device: MyotonPRO

INTERVENTIONS:
Device: MyotonPRO — The MyotonPRO is a non-invasive handheld device that assesses the mechanical and viscoelastic properties of soft tissue (e.g., skin stiffness, elasticity, and relaxation time). In this study, it is used in patients with breast cancer-related lymphedema (BCRL). Each participant is evaluated by two blinded raters to determine intra- and inter-rater reliability.

SUMMARY:
This study aims to evaluate the intra- and inter-rater reliability of the MyotonPRO, a handheld device that measures the viscoelastic properties of the skin, in patients with breast cancer-related lymphedema. Twenty women with unilateral upper extremity lymphedema will be included. Each participant will undergo repeated skin assessments using the MyotonPRO by two independent raters. Additionally, ultrasonographic tissue characteristics and limb volume measurements will be performed. The findings are expected to contribute to the validation of the MyotonPRO for use in clinical lymphedema evaluation.

DETAILED DESCRIPTION:
The study will be conducted at a single center with 20 women diagnosed with unilateral upper extremity lymphedema after mastectomy. Participants will be evaluated using the MyotonPRO device by two trained raters to assess intra- and inter-rater reliability. Ultrasonographic grading of subcutaneous echogenicity and echo-free space, as well as circumference and volume measurements, will be conducted to explore correlations with biomechanical tissue properties. Statistical analysis will include intraclass correlation coefficient (ICC) for reliability and Pearson correlation for validity. This study is expected to support the clinical use of MyotonPRO in lymphedema assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-80 years
* Unilateral upper extremity lymphedema secondary to breast cancer surgery
* Diagnosed with lymphedema at International Society of Lymphology (ISL) Stage 0, I, II, or III
* Willing and able to provide informed consent

Exclusion Criteria:

* Bilateral upper extremity lymphedema
* Cognitive or mental disorders that interfere with cooperation
* Neurological diseases
* Active infection
* Scleroderma or other skin disorders affecting elasticity
* Significant cardiac conditions that may interfere with assessment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Intra- and Inter-Rater Reliability of MyotonPRO Measurements | Within 1 day
  The reliability of the MyotonPRO device will be evaluated through repeated measurements of skin stiffness parameters by two independent raters on the same day. The primary outcome is the intraclass correlation coefficient (ICC) for intra- and inter-rater agreement.
Intra- and Inter-Rater Reliability of MyotonPRO Measurements | Within 1 day
  The reliability of the MyotonPRO device will be evaluated through repeated measurements of skin stiffness parameters by two independent raters on the same day. The primary outcome is the ICC, which quantifies intra- and inter-rater agreement in repeated biomechanical measurements.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality concerns and institutional data protection policies. The study does not include a plan for secondary data analysis or external data use.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30570358/